CLINICAL TRIAL: NCT05033951
Title: Optimizing INITIation of Non-invasive Ventilation in ALS Patients
Acronym: INITIALS
Status: Recruiting | Type: Observational
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, Peter Wijkstra, Prof. Dr. P.J. Wijkstra, University Medical Center Groningen
Other Study IDs: 202000124
Record Dates: First submitted 2021-07-07; First posted 2021-09-05 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: Noninvasive ventilation; Quality of life
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — Standard of Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 42 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort 1: Patients who start NIV in the first two months after the first visit to the HMV
  Interventions: Other: Standard care
- Cohort 2: Patients who do not start NIV in the first two months after the first visit to the HMV.
  Interventions: Other: Standard care

INTERVENTIONS:
Other: Standard care — Both groups: standard care+ questionnaires

SUMMARY:
Objective: The primary objective in this study is to identify which (pheno)type of ALS patient has the most benefit from NIV in improving quality of life.

Study population: Adult patients with ALS, PLS (Primary Lateral Sclerosis) of PSMA (Progressive Spinal Muscular Atrophy) in the Netherlands. Patients will be included during their first visit to one of the HMV centres in the Netherlands.

Main study parameters/endpoints: The main study parameter is change in Quality of Life (QoL) defined as change in ALS Assessment Questionnaire (ALSAQ-40) in patients with ALS after initiation of NIV.

Design: Multi-centre prospective cohort study consisting of 2 non-randomized cohorts, i.e. ALS patients who start NIV and ALS patients who do not start NIV at the time of inclusion in the present study.

Duration: The total duration of the study: 3,5 years. Inclusion period: 30 months. Follow up time after initiation of NIV: 9 months. Thereafter, 6 months will be used for data analysis.

Setting: Involvement of all (4) HMV centres in the Netherlands (Groningen, Maastricht, Rotterdam, Utrecht).

Procedure: 250 ALS patients will be included. During the first regular visit to the HMV centre patients will be asked to participate in the study. Data will be recorded during regular visits to the HMV centre.

DETAILED DESCRIPTION:
First visit:

After informed consent the following data which are gathered as parts of usual care will be recorded in the case report form (CRF):

* Pulmonary function:

  * FVC ( % predicted) upright and supine
  * capillary blood gas analysis, room air (pH, pCO2, HCO3-, pO2)
  * anamnestic questions (Borg scale 0-4)
* Gender
* Age
* Percutaneous Endoscopic Gastrostomy (PEG)/ Percutaneous Radiological Gastrostomy (PRG) tube: yes/no
* Medication
* Weight/ BMI
* Living situation
* Civil status
* The following clinical characteristics from their medical record (from neurologist or rehabilitation specialist):

  * Date of diagnosis
  * Type of ALS at onset
  * ALSFRS-R at the time of diagnosis
  * Pulmonary function at the time of diagnosis
  * Cognitive status (ECAS, ALS-FTD-Q)
  * Medical history
* Validated questionnaires (online):

  * Quality of life questionnaires (SF 36, ALSAQ-40)
  * Respiratory insufficiency questionnaire (SRI)
  * ALS FRS R (patient version)
  * Bulbar symptoms questionnaire (CNS BFS)

After the first visit patients will participate in one of the two cohorts (non-randomized):

* Cohort 1: patients who start NIV in the first two months after the first visit to the HMV
* Cohort 2: patients who do not start NIV in the first two months after the first visit to the HMV.

Cohort 1:

Data will be recorded at the moment of initiation of NIV and 3, 6 and 9 months after initiation. Data will be recorded during regular visits (to the HMV centre or at the patients home).

* Pulmonary function:

  * capillary blood gas, room air (pH, pCO2 (kPa/ mmHg), HCO3- (mmol/l), SaO2 (%))
  * anamnestic questions (Borg scale 0-4)
  * Nocturnal gas exchange by transcutaneous measurement, at the patients home - Mean tcpCO2 (kPa), Maximal tcpCO2 (kPa), mean oxygen saturation (%), lowest oxygen saturation (%)
* Data from NIV equipment (compliance, modus, IPPA, EPAP, freq, mask type)
* Use of NIV

  * hours a day/night
  * In case of no use: why not?
* PEG/ PRG tube: yes/no
* Survival
* Tracheostomy or not
* Weight
* Validated online questionnaires:

  * Quality of life questionnaires (SF 36, ALSAQ-40)
  * Respiratory insufficiency questionnaire (SRI)
  * ALS FRS R (patient version)
  * Bulbar symptoms questionnaire (CNS BFS)
* Nocturnal gas exchange, transcutaneous, at the patients home

Cohort 2:

Data will be recorded every 3 months until initiation of NIV or death or max 1,5 years after the first visit to the HMV.

Data will be recorded during regular visits (to the HMV centre or at the patients home).

* Pulmonary function:

  * Capillary blood gas (pH, pCO2 (kPa/ mmHg), HCO3- (mmol/l), SaO2 (%))
  * anamnestic questions (Borg scale 0-4)
  * Nocturnal gas exchange by transcutaneous measurement, at the patients home - tcpCO2 (kPa), Maximal tcpCO2 (kPa), oxygen saturation (%), lowest oxygen saturation (%)
* PEG/ PRG tube: yes/no
* Survival
* Tracheostomy or not
* Weight
* Cognitive status (from medical record)
* Reason for not starting NIV
* Validated online questionnaires:

  * Quality of life questionnaires (SF 36, ALSAQ-40)
  * Respiratory insufficiency questionnaire (SRI)
  * ALS FRS R (patient version)
  * Bulbar symptoms questionnaire (CNS BFS)
* Nocturnal gas exchange, transcutaneous, at the patients home

If a patient in cohort 2 will start with NIV, the patient will be transferred to cohort 1.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Diagnosis of ALS, PLS or PSMA
* Ability to give informed consent.
* Ability to fill in the questionnaires independently or with assistance of a caregiver.

Exclusion Criteria:

* Use of NIV or invasive ventilation (tracheostomy) at time of first visit to a HMV centre.
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients must be diagnosed with Amyotrophic Lateral Sclerosis (ALS), Progressive Spinal Muscular Atrophy (PSMA) or Primary Lateral Sclerosis (PLS) by a neurologist.
  The patients will be included (after signing informed consent) during the first visit to one of the HMV centres in the Netherlands. Patients must to be able to participate and at least 18 years old
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Health related Quality of Life in patients with ALS | 15 months
  Assessed by Amyotrophic Lateral Sclerosis Assessment Questionnaire (ALSAQ-40) Min score: 0 Max score: 160 Higher scores mean a worse outcome

SECONDARY OUTCOMES:
Survival | 15 months
  Determine the effect of NIV on survival in patients with different ALS phenotypes.
Overall function | 15 months
  Overall function decline based on the ALS Functional Rating Scale Revised (ALS-FRS-R).
  Min score: 0 Max score: 48 Higher scores mean a worse outcome
Forced vital capacity | 15 months
  Pulmonary function based on FVC Min score: 0% Max score: 100% Lower scores mean a worse outcome
Carbondioxide | 15 months
  Pulmonary function based on carbondioxide pCO2 in capillary bloodgas Min score: 4 kPa Max score: 9 kPa Higher score means a worse outcome
Anamnestic questions | 15 months
  Pulmonary function based on anamnestic questions, Borg scale Min score: 0 Max score: 40 Higher score means a worse outcome
Bulbar function | 15 months
  Bulbar function based on questionnaire Center for Neurological Study Bulbar Functional Scale (CNS BFS).
  Min score: 21 Max score: 105 Higher scores means a worse outcome
Weight | 15 months
  Weight in kg Min score: 40 Max score 130 Lower scores mean a worse outcome
General health Quality of Life in patients with severe respiratory insufficiency | 15 months
  Assessed by severe respiratory insufficiency questionnaire (SRI) Min score: 49 Max score: 245 Higher scores mean worse outcome
General health Quality of Life | 15 months
  Assessed by in Short Form Health Survey (SF-36) Min score: 45 Max score: 198 Higher score means a worse outcome

CONTACTS AND LOCATIONS:
Locations (1):
- University medical centre Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No